CLINICAL TRIAL: NCT04481776
Title: Effect of Daily Breakfast Omission Versus Breakfast Consumption on Physical Activity Energy Expenditure and Energy Intake in Adolescent Girls Who Habitually Skip Breakfast: a 7-day Crossover Trial
Brief Title: Breakfast Omission and Energy Balance in Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Dr Julia Fruer, Senior Lecturer in Health, Nutrition and Exercise, University of Bedfordshire
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Bedfordshire
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Adolescent Obesity; Insulin Resistance; Adolescent Behavior
Keywords: Breakfast; Physical activity; Nutrition; Appetite; Sedentary
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Adolescent Behavior; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast consumption (Experimental): Participants will be asked to consume a standardised breakfast at home before 09:00 for seven consecutive days. The energy content of the breakfast will be 25% of individual measured resting metabolic rate. Prior to the experimental conditions, the participants will select one wholegrain, high-fibre ready-to-eat cereals (with the option of adding raisins) and fruit juice from a limited selection. Thus, breakfast composition will be controlled within participants, but not between participants to account for individual preferences. To ensure that the correct amount of each breakfast item is consumed, food items will be provided to the participants in pre-packaged containers and the participants will be provided with a marked beaker to measure their milk and juice each morning. The only exception is that parents will be asked to provide the 1.8% milk.
  Interventions: Other: Breakfast consumption
- Breakfast omission (Experimental): Participants were asked to abstain from all energy-providing nutrients before 10:30 for seven consecutive days.
  Interventions: Other: Breakfast omission

INTERVENTIONS:
Other: Breakfast consumption — Standardised breakfast consumption across seven days
  Arms: Breakfast consumption
Other: Breakfast omission — No breakfast consumed across seven days
  Arms: Breakfast omission

SUMMARY:
There is a distinct lack of experimental evidence on whether breakfast consumption and omission affect energy balance-related variables. This research is of particular relevance to adolescent girls due to concerns of low rates of breakfast consumption and physical activity in this population. This study aims to compare the effect of seven consecutive days of breakfast omission with standardised breakfast consumption on free-living physical activity energy expenditure, energy intake and perceived appetite and energy levels in adolescent girls.

DETAILED DESCRIPTION:
Observational reports showing infrequent breakfast consumption to be associated with increased adiposity and cardiometabolic disease risk in children and adolescents have fuelled concerns over the low prevalence of habitual breakfast consumption among adolescents. Yet, only experimental study designs can determine the causal effects of breakfast consumption on health-related variables and such research has typically targeted adults. Adolescent girls may respond differently to manipulations in breakfast consumption than adults because they have distinct hormonal, metabolic and behavioural profiles. Further, a link between breakfast and physical activity in adolescent girls has particular public health relevance because the adolescent decline in both breakfast consumption frequency and physical activity is more pronounced in girls than in boys. Thus, the primary aim of the current study is to use a randomised, cross-over design to compare the effect of seven consecutive days of breakfast omission with standardised breakfast consumption on free-living PAEE in adolescent girls. The secondary aims are to examine the effects on energy intake, perceived appetite and energy levels.

Using a randomized crossover design, girls aged 11-14 years will complete two, 7-day conditions. A standardized breakfast will consumed every day before 09:00 in the daily breakfast consumption condition. No energy-providing nutrients will consumed (i.e., only water) before 10:30 in the breakfast omission condition. Combined heart rate-accelerometry will be used to estimate physical activity energy expenditure and digital photography complemented with written food diaries will be used to assess energy intake during each condition; these data will be separated into three time segments: wake to 10:30, 10:30 to 15:30 and 15:30 to bed. Visual analogue scales will be used to assess perceptions of hunger, fullness, tiredness and energy levels on waking and at 09:00 and 10:30. Statistical analyses will be completed using condition by time of day linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Parental informed consent
* Child assent

Exclusion Criteria:

* Health related issues identified from a health screen questionnaire that could be adversely affected by participation or could affect the study outcomes (e.g., allergies to the breakfast meals, fitted with a pacemaker)
* Unable to walk or wear a combined heart rate-accelerometer on the chest.

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Physical activity energy expenditure (kJ/day) | Seven days
  Free-living physical activity energy expenditure from sedentary, light, moderate and vigorous activities (kJ/day) assessed using combined heart rate-accelerometry across seven consecutive days.
Time spent in physical activity (minutes/day) | Seven days
  Time spent sedentary and in light, moderate and vigorous physical activity (minutes/day) assessed using combined heart rate-accelerometry across seven consecutive days.

SECONDARY OUTCOMES:
Energy intake (kJ/day) | Four days
  Energy intake (kJ/day) assessed using combined digital photography and food diaries across four days.
Carbohydrate intake (g/day) | Four days
  Carbohydrate intake (g/day) assessed using combined digital photography and food diaries across four days.
Fat intake (g/day) | Four days
  Fat intake (g/day) assessed using combined digital photography and food diaries across four days.
Protein intake (g/day) | Four days
  Protein intake (g/day) assessed using combined digital photography and food diaries across four days.
Fibre intake (g/day) | Four days
  Fibre intake (g/day) assessed using combined digital photography and food diaries across four days.
Perceived hunger (mm) | Four days
  Perceived hunger (mm) assessed using 0-100 mm visual analogue scales on waking, at 09:00 and at 10:30 on four days. Higher values equate to higher hunger.
Perceived fullness (mm) | Four days
  Perceived fullness (mm) assessed using 0-100 mm visual analogue scales on waking, at 09:00 and at 10:30 on four days. Higher values equate to higher fullness.
Perceived tiredness levels (mm) | Four days
  Perceived tiredness levels (mm) assessed using 0-100 mm visual analogue scales on waking, at 09:00 and at 10:30 on four days. Higher values equate to higher tiredness.
Perceived energy levels (mm) | Four days
  Perceived energy levels (mm) assessed using 0-100 mm visual analogue scales on waking, at 09:00 and at 10:30 on four days. Higher values equate to higher energy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Julia K Fruer, PhD, Principal Investigator — University of Bedfordshire
Locations (1):
- University of Bedfordshire, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No